CLINICAL TRIAL: NCT04064957
Title: Hope Biosciences Autologous Adipose-derived Mesenchymal Stem Cell Therapy for Chronic Spinal Cord Injury (HBSCI02), Individual Patient Expanded Access IND to Evaluate the Safety and Efficacy of HB-adMSCs for the Treatment of Spinal Cord Injury (HBSCI04 & HBSCI05)
Brief Title: Individual Patient Expanded Access IND of Hope Biosciences Autologous Adipose-derived Mesenchymal Stem Cells for Spinal Cord Injury
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBSCI02, HBSCI04, HBSCI05
Record Dates: First submitted 2019-08-19; First posted 2019-08-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; MSCs; HB-adMSCs; chronic SCI; stem cells; autologous
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: HB-adMSCs
  Other Names: Hope Biosciences autologous adipose-derived mesenchymal stem cells

SUMMARY:
HBSCI02:

This protocol is part of an FDA Individual Patient Non-emergency Expanded Access Request submitted on behalf of a 38-year-old father and husband who on August 4, 2017 at about 4:30pm, slipped off a boat head-first while in the Florida Keys for a family wedding, and was immediately unable to move his legs. He discharged to Texas via air ambulance for physical rehabilitation on August 23, 2017 with a diagnosis of ASIA B (American Spinal Injury Association) C-5 SCI (spinal cord injury).

HBSCI04:

This Individual Patient Expanded Access IND has been created per the request of a 75-year-old man who has been diagnosed with Spinal Cord Injury. The patient requested this Expanded Access IND with the purpose of possible restoration of nerve transmission and restoring sensation in his upper and lower body using intravenous autologous adipose derived mesenchymal stem cells.

HBSCI05:

This Individual Patient Expanded Access IND has been created per the request of a 26-year-old man who has been diagnosed with Spinal Cord Injury. The patient is a 26-year-old male who suffered an unstable C-6 compressive fracture, crushing the vertebral body and retropulsion of a large bone fragment into the vertebral canal, stenosing 75% of spinal canal in a diving accident on 12/4/2021 in Belize City, Belize. The injury classification is C-6 Asia A injury. The injury left him with flaccid paralysis below the level of C-7 dermatome.

DETAILED DESCRIPTION:
HBSCI02:

Once the eligibility is confirmed, approximately 1-3 weeks after the screening/baseline visit, the subject will receive the first infusion. Subsequent treatments will occur every other week in the subject's home, administered by a nurse.

On each of these visits, the subject will receive one autologous HB-adMSC infusion of 200 million (2 x 10^8 cells) total cells. Every infusion visit will include the following procedures:

1. Interval H&P and concomitant medications update.
2. QOL and Disability (SCIM self eval) surveys will be completed by the subject with the assistance of the primary caregiver.
3. Vital signs monitoring will be initiated (Heart Rate, BP, Resp., Temp., SpO2).
4. A peripheral IV line will be inserted.
5. A blood sample for clinical labs will be drawn monthly during the infusion period.
6. A "time out" verification of patient/consent/procedure/cell product will be performed.
7. The HB-adMSC infusion will be given by through the peripheral IV.
8. Assessment for Infusion Related AE/SAEs.
9. The subject will be monitored for a minimum of 2 hours.

In-Person Visits The subject will return to the Clinical Trial Network CTN site for In-Person visits to occur at Screening, Baseline and Week twelve (12), twenty-six (26) and at Week fifty-two (52). Week 52 visit will serve as the End of Study visit. The end of study (EOS) visit will include an MRI of the c-spine as well as all of the study procedures for Follow-up Visits without Infusion. A written summary of the results of the treatment, including adverse events will be submitted to the FDA after completion of the last follow-up visit.

Visits without infusion will include:

1. Interval H&P and concomitant medications update.
2. QOL and Disability (SCIM self eval) surveys will be completed by the subject with the assistance of the primary caregiver.
3. Vital signs monitoring will be initiated (Heart Rate, BP, Resp., Temp., SpO2),
4. A Physical and Neuro Exam (Asia Impairment Scale) will be completed
5. A blood sample for clinical labs (CBC with Platelets, CMP, PT, PTT, TNFa, IL6, CRP) will be drawn.
6. Video documentation of patient condition.
7. Assessment for infusion related AEs/SAEs
8. Weight

HBSCI04:

This expanded access IND was created at the request of the subject who already has his own stem cells banked at Hope Biosciences, LLC. After receiving authorization from FDA and Western IRB, the subject will be contacted and provided with a copy of the informed consent for review. If consent is obtained, the principal investigator or delegated staff will collect patient's medical history and schedule the date for the Infusion 1.

The informed consent process will be documented in the subject's record and will include the discussion points mentioned above. A copy of the signed informed consent will be given to the patient and also placed in the record.

Subject will receive a total of fourteen autologous HB-adMSCs infusion of 200 million cells with a dosing interval of approximately 2 weeks for the first five infusions and 28 days for the remaining 9 infusions over a 44-week period, Laboratory assessments will be collected at Infusion 1, 10, and EOS.

Other assessments should be completed during these visits by the Principal Investigator and/or delegated staff in order to evaluate the safety and efficacy of HB-adMSCs.

1. Collection of Medical History.
2. Collection of Concomitant Medications.
3. Collection of Vital Signs (Respiratory Rate, Blood Pressure, Body Temperature, Heart Rate and Oxygen Saturation). Vital Signs will be collected for 2 hours post investigational product exposure. Every 15 minutes for the first hour and every 30 minutes after that. If it is indicated by principal investigator vital signs should be collected more frequently.
4. EMG NCV is required to be completed at Infusion 1 and EOS. If an EMG NCV has not been done within 28 days of these visits, the Principal Investigator will place an order to obtain it. Any EMG NCV done within 28 days of the visit as standard of care can be used for this requirement.
5. A Physical and Neuro Examination will be completed by the principal investigator.
6. Neuro QOL Scale at Infusion 1, 5, 7, 9, 11 and 13.
7. SCIM (Spinal Cord Independence Measure) Clinician assessment at Infusion 1, 10 and EOS.
8. SCIM (Self-Assessment) at Infusion 1, 10, and EOS.
9. A video documentation of the subject will be recorded during Infusion 1 with the purpose of observing his general physical health, trunk stability and if there are other new changes.
10. Laboratory Samples. A blood sample for clinical labs - CBC with Platelets, CMP, PT, PTT, INR, as well as C-reactive protein and Sedimentation rate to be collected at Infusion 1 and 10 and EOS.
11. Telephone Encounter 24 hours after each infusion to evaluate the incidence of any Adverse event or Serious Adverse Events.

Follow Up Week 48 Phone Call

1. Update medical history and concomitant medications if there is any new information.
2. Assess the incidence of any Adverse event or Serious Adverse Events since last infusion.

End of Study End of Study will include the following study procedures,

1. Interval H&P and concomitant medications update.
2. Neuro QOL and Disability (SCIM self eval) surveys will be completed by the subject.
3. EMG NCV is required to be completed at this visit. If an EMG NCV has not been done within 28 days of this visit, the Principal Investigator will place an order to obtain it. Any EMG NCV done within 28 days of the visit as standard of care can be used for this requirement.
4. Vital signs monitoring will be initiated (Heart Rate, Blood Pressure, Resp., Temp., SpO2)
5. A Physical and Neuro Examination will be completed by the principal investigator.
6. A blood sample for clinical labs will be collected CBC with Platelets, CMP, PT, PTT, INR, as well as C-reactive protein and Sedimentation rate.
7. A video documentation of the subject will be recorded during this visit with the purpose of observing his general physical health and if there are other new changes.
8. Assess the incidence of any Adverse event or Serious Adverse Events since last infusion.

HBSCI05:

This expanded access IND was created at the request of the subject who already has his own stem cells banked at Hope Biosciences, LLC. After receiving authorization from FDA and Western IRB, the subject will be contacted and provided with a copy of the informed consent for review. The Principal Investigator or delegated staff will contact the patient by telephone and explain the study procedures (including cell infusion, and safety assessment procedures), follow-up visits, potential risks and benefits of the study, alternatives, and the voluntary nature of participation.

Ample time will be given for the patient to ask questions and make a decision about participation. If consent is obtained, the principal investigator or delegated staff will collect patient's medical history and schedule the date for the Infusion 1.

The informed consent process will be documented in the subject's record and will include the discussion points mentioned above. A copy of the signed informed consent will be given to the patient and also placed in the record.

Subject will receive a total of fourteen autologous HB-adMSCs infusion of 200 million cells with a dosing interval of approximately 2 weeks for the first five infusions and 28 days for the remaining 9 infusions over a 44-week period, volume to administer 250 ml of Sodium Chloride 0.9% and infusion rate 4 - 5 ml/min. Laboratory assessments will be collected at Infusion 1, 10, and EOS.

Other assessments should be completed during these visits by the Principal Investigator and/or delegated staff in order to evaluate the safety and efficacy of HB-adMSCs.

1. Collection of Medical History.
2. Collection of Concomitant Medications.
3. Collection of Vital Signs (Respiratory Rate, Blood Pressure, Body Temperature, Heart Rate and Oxygen Saturation). Vital signs will be taken for 1 hour during exposure to the research product with an interval of 15 minutes. However, if warranted or indicated by the investigator vital signs will be taken more frequently or longer if necessary.
4. EMG NCV is required to be completed at Infusion 1 and EOS. If an EMG NCV has not been done within 28 days of these visits, the Principal Investigator will place an order to obtain it. Any EMG NCV done within 28 days of the visit as standard of care can be used for this requirement.
5. A Physical and Neuro Examination will be completed by the principal investigator.
6. Neuro QOL Scale at Infusion 1, 5, 7, 10, 11 and 13, and EOS.
7. SCIM (Spinal Cord Independence Measure) Clinician assessment at Infusion 1, 10 and EOS.
8. SCIM (Self-Assessment) at Infusion 1, 10, and EOS.
9. A video documentation of the subject will be recorded during Infusion 1 with the purpose of observing his general physical health, trunk stability and if there are other new changes.
10. Laboratory Samples. A blood sample for clinical labs - CBC with Platelets, CMP, PT, PTT, INR, as well as C-reactive protein and Sedimentation rate to be collected at Infusion 1 and 10 and EOS.
11. Telephone Encounter 24 hours after each infusion to evaluate the incidence of any Adverse event or Serious Adverse Events.

Follow Up Week 48 Phone Call

1. Update medical history and concomitant medications if there is any new information.
2. Assess the incidence of any Adverse event or Serious Adverse Events since last infusion.

End of Study

End of Study will include the following study procedures,

1. Interval H&P and concomitant medications update.
2. Neuro QOL and Disability (SCIM self eval) surveys will be completed by the subject.
3. EMG NCV is required to be completed at this visit. If an EMG NCV has not been done within 28 days of this visit, the Principal Investigator will place an order to obtain it. Any EMG NCV done within 28 days of the visit as standard of care can be used for this requirement.
4. Vital signs monitoring will be initiated (Heart Rate, Blood Pressure, Resp., Temp., SpO2)
5. A Physical and Neuro Examination will be completed by the principal investigator.
6. A blood sample for clinical labs will be collected CBC with Platelets, CMP, PT, PTT, INR, as well as C-reactive protein and Sedimentation rate.
7. A video documentation of the subject will be recorded during this visit with the purpose of observing his general physical health and if there are other new changes.
8. Assess the incidence of any Adverse event or Serious Adverse Events since last infusion.

ELIGIBILITY:
HBSCI02:

Inclusion Criteria:

1. Adult individual 18 yr. of age or older.
2. Cognitively intact and capable of giving informed consent.
3. Clinical diagnosis of a non-penetrating traumatic SCI to the cervical spine
4. Patient and Caregiver agree to use Care Connect app or web version of VirTrial platform for virtual visits.

Exclusion Criteria:

1. Prior history of:

   1. Recent or ongoing infection,
   2. Clinically significant cardiovascular, lung, renal, hepatic, or endocrine disease,
   3. Neurodegenerative disorders,
   4. Cancer,
   5. Immunosuppression as defined by WBC < 3, 000 cells/ml at baseline screening,
   6. Chemical or ETOH dependency,
2. Having a contraindication to MRI scans
3. Other acute or chronic medical conditions that, in the opinion of the investigator, may increase the risks associated with study participation or HB-adMSC administration
4. Participation in other interventional research studies.
5. Unwillingness to return for follow-up visits

HBSCI04:

Inclusion Criteria:

1. Adult individual 18 years of age or older.
2. Cognitively intact and capable of giving informed consent.
3. Clinical diagnosis of Spinal Cord Injury.
4. Subject has mesenchymal stem cells banked at Hope Biosciences.
5. The patient accepts to receive treatment and to comply with follow-up visits.

Exclusion Criteria:

1. Clinically significant, uncontrolled cardiovascular, lung, renal, hepatic, or endocrine disease or any other acute or chronic medical condition that, in the opinion of the investigator may increase the risks associated with study participation.
2. Active Alcohol or Drug addiction.
3. Participation in concurrent interventional research studies during this study.
4. Severe organ failure (heart, kidney or liver) confirmed by additional tests or medical history.
5. Unwillingness to return for follow-up visits.

HBSCI05:

Inclusion Criteria:

1. Adult individual 18 years of age or older.
2. Cognitively intact and capable of giving informed consent.
3. Clinical diagnosis of Spinal Cord Injury.
4. Subject has mesenchymal stem cells banked at Hope Biosciences.
5. The patient accepts to receive treatment and to comply with follow-up visits.

Exclusion Criteria:

1. Clinically significant, uncontrolled cardiovascular, lung, renal, hepatic, or endocrine disease or any other acute or chronic medical condition that, in the opinion of the investigator may increase the risks associated with study participation.
2. Active Alcohol or Drug addiction.
3. Participation in concurrent interventional research studies during this study.
4. Severe organ failure (heart, kidney or liver) confirmed by additional tests or medical history.
5. Unwillingness to return for follow-up visits.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Djamchid Lotfi, MD, Principal Investigator — Hope Biosciences Stem Cell Research Foundation
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States

REFERENCES:
- See also: Hope Biosciences — http://www.hope.bio
- See also: Hope Biosciences Stem Cell Research Foundation — https://www.hopebio.org/